CLINICAL TRIAL: NCT04683055
Title: Phacoemulsification Combined With Trabeculectomy Versus Phacoemulsification Combined With Trabeculotomy for Treatment of Chronic Angle Closure Glaucoma
Brief Title: Phaco-Trabeculotomy Vs Phaco-Trabeculectomy
Acronym: PDT vs PT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud F. Rateb, Assitant Professor of Ophthalmology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB17300506
Record Dates: First submitted 2020-12-20; First posted 2020-12-24 (Actual); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: Ophthalmopathy; Glaucoma; Glaucoma, Angle-Closure
MeSH Terms: conditions — Eye Diseases; Glaucoma; Glaucoma, Angle-Closure | interventions — Trabeculectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phacoemulsification combined with trabeculectomy (Active Comparator): Patients will undergo Two site phacoemulsification combined with trabeculectomy with Mitomycin C
  Interventions: Procedure: Phacoemulsification combined with trabeculectomy
- Phacoemulsificaiton combined with ab-externo trabeculotomy (Active Comparator): Patients will undergo two phacoemulsification combined with deep sclerectomy and ab-externo trabeculotomy
  Interventions: Procedure: Phacoemulsificaiton combined with ab-externo trabeculotomy

INTERVENTIONS:
Procedure: Phacoemulsification combined with trabeculectomy — Patients with chronic angle closure glaucoma assigned to this group will have fornex based trabeculectomy at superior limbus and then phacoemulsification via temporal incision
  Arms: Phacoemulsification combined with trabeculectomy
Procedure: Phacoemulsificaiton combined with ab-externo trabeculotomy — Patients with chronic angle closure glaucoma assigned to this group will have Deep Sclerectomy with ab externo trabeculotomy at superior limbus and then phacoemulsification via temporal incision
  Arms: Phacoemulsificaiton combined with ab-externo trabeculotomy

SUMMARY:
A prospective, randomized comparative study on adult patients with synechial angle closure glaucoma.

DETAILED DESCRIPTION:
Patients were randomized into two groups: group A : patients will undergo two site phacoemulfication combined with trabeculectomy Group B with Phacoemulsification combined with ab-externo trabeculotomy. Preoperative assessments including full ophthalmic examination, anterior segment Optical Coherence Tomography (OCT) of the angle , endothelial cell count , visual fiend Perimetry and Biometry. Patients were followed up: first day, first week and every two months for 6 month. We will compare adverse effects and outcomes in both groups.

ELIGIBILITY:
Inclusion Criteria:

Patients with chronic angle closure glaucoma, with or without peripheral anterior synechiae, age more than 18

Exclusion Criteria:

* Patient unable for follow up
* Patients with corneal or retinal disease that affects visual outcome of surgery
* Patients with previous glaucoma procedure in the eye of study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Absolute Success | 1,3,6 months
  Reduction of IOP more than 30% on no glaucoma drops
Visual outcome | 1,3,6 month
  Uncorrected visual acuity by Snellen's chart

SECONDARY OUTCOMES:
Adverse events | 1 week, 1 month, 3 months, 6 months
  all intraoperative and postoperative adverse events witt be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data in the study , after completion after de-identification
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after publication and for five years
Access Criteria: Anyone who wants to access data

REFERENCES:
- [Background] Lichter PR, Musch DC, Gillespie BW, Guire KE, Janz NK, Wren PA, Mills RP; CIGTS Study Group. Interim clinical outcomes in the Collaborative Initial Glaucoma Treatment Study comparing initial treatment randomized to medications or surgery. Ophthalmology. 2001 Nov;108(11):1943-53. doi: 10.1016/s0161-6420(01)00873-9. PMID 11713061
- [Background] Rebolleda G, Munoz-Negrete FJ. Phacoemulsification in eyes with functioning filtering blebs: a prospective study. Ophthalmology. 2002 Dec;109(12):2248-55. doi: 10.1016/s0161-6420(02)01246-0. PMID 12466166
- [Background] Hansapinyo L, Choy BNK, Lai JSM, Tham CC. Phacoemulsification Versus Phacotrabeculectomy in Primary Angle-closure Glaucoma With Cataract: Long-Term Clinical Outcomes. J Glaucoma. 2020 Jan;29(1):15-23. doi: 10.1097/IJG.0000000000001397. PMID 31702714
- [Background] Toteberg-Harms M, Wachtl J, Schweier C, Funk J, Kniestedt C. Long-term efficacy of combined phacoemulsification plus trabeculectomy versus phacoemulsification plus excimer laser trabeculotomy. Klin Monbl Augenheilkd. 2017 Apr;234(4):457-463. doi: 10.1055/s-0043-100291. Epub 2017 Mar 6. PMID 28264221